CLINICAL TRIAL: NCT01149993
Title: Attenuating Ischemia Reperfusion Injury After Living Donor Renal Transplantation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA clinical hold, IND withdrawn.
Sponsor: Georgetown University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Keith Melancon,MD, Director of kidney and pancreas transplantation, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-496
Record Dates: First submitted 2010-06-21; First posted 2010-06-24 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Kidney Transplantation; Renal Transplantation; Reperfusion Injury
Keywords: living donation; kidney transplantation; delayed graft function; ischemia reperfusion injury
MeSH Terms: conditions — Reperfusion Injury; Delayed Graft Function | interventions — Mycophenolic Acid; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pre-transplant immunosuppression (Experimental): subjects in this arm will receive Myfortic 720mg twice daily for 7 days prior to transplantation. Intra-operatively, the donor kidney will receive an infusion of Thymoglobulin, prior to the transplantation.
  Interventions: Drug: Myfortic (mycophenolic acid); Drug: Thymoglobulin (anti-thymocyte globulin)
- pre-transplant induction (Experimental): subjects in this arm will not receive any pre-transplant immunosuppression. However, the donor kidney will receive an infusion of Thymoglobulin prior to transplantation.
  Interventions: Drug: Myfortic (mycophenolic acid); Drug: Thymoglobulin (anti-thymocyte globulin)
- standard of care (Active Comparator): subjects in this arm will not receive any pre-transplant immunosuppression, and the donor kidney will not receive an additional dose of Thymoglobulin prior to transplantation. This is the standard of care protocol for Georgetown University Hospital
  Interventions: Drug: Myfortic (mycophenolic acid); Drug: Thymoglobulin (anti-thymocyte globulin)

INTERVENTIONS:
Drug: Myfortic (mycophenolic acid) — 720mg twice a day for 7 days prior to transplantation
  Arms: pre-transplant immunosuppression
Drug: Myfortic (mycophenolic acid) — 720mg twice a day after transplant
Drug: Thymoglobulin (anti-thymocyte globulin) — up to 25 mg will be infused into the renal artery of a donor kidney prior to transplantation into the recipient.
  Arms: pre-transplant immunosuppression; pre-transplant induction
Drug: Thymoglobulin (anti-thymocyte globulin) — standard of care for Georgetown University Hospital: 1.5 mg/kg/day infused over 6 hours.

SUMMARY:
Patients undergoing living donor renal transplant will be asked to participate to determine whether pre-operative dosing of immunosuppressive medication, and the donor organ receiving an additional dose of antibody induction therapy helps to alleviate potential damage to the transplanted organ post-transplant. A number of lab tests will be done post-transplant to determine how well the kidney is functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to provide written informed consent.
2. All recipients of a kidney from a living donor only, either a de novo transplant, or re-transplant
3. All patients evaluated and listed with the United Network for Organ Sharing (UNOS) who are eligible to receive a kidney transplant under GUH's standard protocol.
4. Patients between 18-80 years of age

Exclusion Criteria:

1. Recipients of multi-organ transplant
2. Patients with known allergies of hypersensitivities to any of the drugs used in this protocol
3. Recipients of kidneys from a deceased donor
4. Recipients who are co-infected with Hepatitis B, Hepatitis C or HIV
5. Women who are pregnant
6. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle or sexual orientation precludes intercourse with a male partner unless they agree to avoid pregnancy throughout the duration of the trial and for 3 months following the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
reduction in ischemia reperfusion injury | one year
  Monitor immediate graft functioning, mitochodrial membrane potential, serum creatinine, and cylex immunomonitoring to determine if pre-transplant immunosuppression, and an additional intra-operative dose of induction agent helps to reduce ischemic reperfusion injury.

SECONDARY OUTCOMES:
secondary outcomes | one year
  incidence of acute rejection, graft survival, patient survival, change in cylex values

CONTACTS AND LOCATIONS:
Overall Officials: Joseph K Melancon, MD, Principal Investigator — Georgetown University Hospital